CLINICAL TRIAL: NCT04971226
Title: A Phase III, Multi-center, Open-label, Randomized Study of Oral Asciminib Versus Investigator Selected TKI in Patients With Newly Diagnosed Philadelphia Chromosome Positive Chronic Myelogenous Leukemia in Chronic Phase
Brief Title: A Study of Oral Asciminib Versus Other TKIs in Adult Patients With Newly Diagnosed Ph+ CML-CP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CABL001J12301; 2023-508838-33-00 (Registry Identifier: EU CTIS)
Expanded Access: NCT04360005 (Available)
Record Dates: First submitted 2021-06-08; First posted 2021-07-21 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Myeloid Leukemia (CML) Philadelphia Chromosome Positive
Keywords: Asciminib; Chronic Myeloid Leukemia; CML; Philadelphia Chromosome; TKIs; Bosutinib; Dasatinib; Nilotinib; Imatinib; Treatment-free remission
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Philadelphia Chromosome | interventions — Imatinib Mesylate; nilotinib; bosutinib; Dasatinib; asciminib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Asciminib (Experimental): Patients will take asciminib 80 mg QD under fasting conditions on ongoing basis; Patients will be randomized 1:1 asciminib versus Investigator selected TKIs
  Interventions: Drug: Asciminib
- Investigator selected TKIs (Active Comparator): Patients will take on ongoing basis the Investigator selected TKIs that will include one of the below treatments:
  Imatinib 400 mg QD administered with food Nilotinib 300 mg BID administered under fasting conditions Dasatinib 100 mg QD administered with or without a meal Bosotunib 400 mg QD administered with food
  Interventions: Drug: Imatinib; Drug: Nilotinib; Drug: Bosutinib; Drug: Dasatinib

INTERVENTIONS:
Drug: Imatinib — Comes in 100 mg and 400 mg tablets and taken orally
  Other Names: STI571
  Arms: Investigator selected TKIs
Drug: Nilotinib — Comes in 150 mg and 200 mg capsules and taken orally
  Other Names: AMN107
  Arms: Investigator selected TKIs
Drug: Bosutinib — Comes in 100 mg and 400 mg tablets and taken orally
  Arms: Investigator selected TKIs
Drug: Dasatinib — Comes in 20 mg, 50 mg, 70 mg and 100 mg tablets and taken orally
  Arms: Investigator selected TKIs
Drug: Asciminib — Comes in 40 mg tablets and taken orally
  Other Names: ABL001
  Arms: Asciminib

SUMMARY:
The study is designed to compare the efficacy of asciminib 80 mg QD versus Investigator selected Tyrosine Kinase Inhibitor (TKI) for the treatment of newly diagnosed, previously untreated patients with Ph+ CML-CP. The Investigator selected TKI will be one of the following treatment options for first-line treatment of CML-CP - imatinib 400 mg QD or nilotinib 300 mg BID or dasatinib 100 mg QD or bosutinib 400 mg QD.

This study has three periods: 1. Treatment period for all randomized participants, 2. Optional Treatment-Free Remission (TFR) period only for participants meeting TFR eligibility criteria and 3. Treatment Re-Initiation (TRI) period only for participants who relapsed after TFR attempt.

DETAILED DESCRIPTION:
This study is a phase III, multi-center, open-label, randomized study of oral asciminib 80 mg QD versus Investigator selected TKI (imatinib, nilotinib, dasatinib, or bosutinib) in adult patients with newly diagnosed Ph+ CML-CP. All comparator TKIs will be made available, unless not permitted by local regulations or local Health Authority or not approved for the treatment of CML in the country.

Approximately 402 patients will be randomized in a 1:1 ratio to asciminib and Investigator selected TKI to join the treatment period.

Randomization will be stratified based on the following two stratification factors:

* ELTS score (low versus intermediate versus high)
* Pre-randomization selected TKI (imatinib versus 2G TKI (nilotinib or dasatinib or bosutinib)).

Prior to randomization, the Investigator, in consultation with the patient, considering the current treatment paradigm and patient characteristics and comorbidities, will make a selection of preference for imatinib or 2G TKI (nilotinib or dasatinib or bosutinib) if the patient is randomized to the comparator arm. The stratified randomization based on these two stratification factors will help to achieve a balance across the treatment arms for the possible comorbidities and baseline characteristics of patients enrolled in the study.

To further ensure that the distribution of patients, between imatinib and 2G TKIs (nilotinib or dasatinib or bosutinib), in the Investigator selected TKI arm is reflective of the use of these agents in clinical practice, the enrollment into the strata of imatinib versus 2G TKI (nilotinib or dasatinib or bosutinib) based on the pre-randomization selection of TKI will be managed by Interactive Response Technology to be approximately 50% versus 50%.

Treatment arms: The study will have 2 treatment arms:

* Arm 1: asciminib 80 mg QD under fasting conditions
* Arm 2: Investigator selected TKI that will include one of the below treatments:
* Imatinib 400 mg QD administered with food
* Nilotinib 300 mg BID administered under fasting conditions
* Dasatinib 100 mg QD administered with or without meal
* Bosutinib 400 mg QD administered with food.

Apart from the treatment period described above, the present study comprises an optional Treatment-Free Remission (TFR) Period enrolling consenting participants of the treatment period (receiving asciminib or IS-TKI) who will discontinue their randomized treatment if they meet per protocol eligibility criteria. The optional TFR Period will last at least 2 years to assess the feasibility of TFR and TFR outcomes following discontinuation of their randomized treatment (asciminib or IS-TKI).

In addition, during the TFR Period, participants who will lose major molecular response (MMR) must re-initiate treatment and will enter into a Treatment Reinitiation (TRI) Period.

During the treatment period, no crossover of study treatment across arms and no change of study treatment within the Investigator selected TKI will be allowed. For specifically participants who must transition into the TRI Period, at the time of treatment re-initiation: a) participants who were previously treated with asciminib will resume asciminib at the same dose prior to entry into TFR. b) participants who were on IS-TKI may either continue with the same study treatment they were randomized to and at the same dose prior to entry into TFR or may switch to asciminib with a starting dose of 80 mg QD.

Duration of Study treatment: Patients on the study will continue to receive the assigned treatment until the End of Study, premature discontinuation due to treatment failure, disease progression or intolerance, due to Investigator or participant decision. or due to patient going to TFR Period and/or TRI Period.

Duration of study: The End of Study will occur 8 years from the last patient first treatment in the study. Patients who discontinue study treatment prematurely due to any reason, will be followed up for survival and progression (to AP/BC) until the End of Study.

ELIGIBILITY:
Inclusion Criteria for treatment period:

Participants eligible for inclusion in this study must meet all of the following criteria:

* Male or female patients ≥ 18 years of age.
* Participants with CML-CP within 3 months of diagnosis.
* Diagnosis of CML-CP (ELN 2020 criteria) with cytogenetic confirmation of Philadelphia chromosome

Documented chronic phase CML will meet all the below criteria (Hochhaus et al 2020):

* < 15% blasts in peripheral blood and bone marrow,
* < 30% blasts plus promyelocytes in peripheral blood and bone marrow,
* < 20% basophils in the peripheral blood,
* Platelet count ≥ 100 x 10^9/L (≥ 100,000/mm^3),
* No evidence of extramedullary leukemic involvement, with the exception of hepatosplenomegaly.

  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  * Adequate end organ function as defined by:
* Total bilirubin < 3 x ULN; patients with Gilbert's syndrome may only be included if total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤ 1.5 x ULN
* Creatinine clearance (CrCl) ≥ 30 mL/min as calculated using Cockcroft-Gault formula,
* Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN - ≤ 1.5 x ULN, value must be considered not clinically significant and not associated with risk factors for acute pancreatitis

  - Participants must have the following laboratory values within normal limits or corrected to within normal limits with supplements prior to randomization:
* Potassium (potassium increase of up to 6.0 mmol/L is acceptable if associated with CrCl* ≥ 90 mL/min)
* Total calcium (corrected for serum albumin); (calcium increase of up to 12.5 mg/dl or 3.1 mmol/L is acceptable if associated with CrCl* ≥ 90 mL/min)
* Magnesium (magnesium increase of up to 3.0 mg/dL or 1.23 mmol/L if associated with CrCl* ≥ 90 mL/min)
* For patients with mild to moderate renal impairment (CrCl* ≥ 30 mL/min and <90 mL/min) - potassium, total calcium (corrected for serum albumin) and magnesium should be ≥ LLN or corrected to within normal limits with supplements prior to randomization.
* *CrCl as calculated using Cockcroft-Gault formula

  * Ability to provide written informed consent prior to any study related screening procedures being performed.
  * Evidence of typical BCR-ABL1 transcript [e14a2 and/or e13a2] at the time of screening which is amenable to standardized Real time quantitative polymerase chain reaction (RQ-PCR) quantification.

Exclusion Criteria for Treatment period:

* Previous treatment of CML with any other anticancer agents including chemotherapy and/or biologic agents or prior stem cell transplant, with the exception of hydroxyurea and/or anagrelide. Treatment with either imatinib, or nilotinib, or dasatinib or bosutinib for ≤2 weeks is allowed, but no other treatment with other tyrosine kinase inhibitors prior to randomization is permitted.
* Known cytopathologically confirmed CNS infiltration (in absence of suspicion of CNS involvement, lumbar puncture not required).
* Impaired cardiac function or cardiac repolarization abnormality including but not limited to any one of the following:

  * History within 6 months prior to starting study treatment of myocardial infarction (MI), angina pectoris, coronary artery bypass graft (CABG)
  * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g., bifascicular block, Mobitz type II and third degree AV block)
  * QTc ≥ 450 ms (male patients), ≥460 ms (female patients) on the average of three serial baseline ECG (using the QTcF formula) as determined by central reading. If QTcF ≥ 450 ms and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc.
  * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
  * Risk factors for Torsades de Pointes (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia
  * Concomitant medication(s) with a "Known risk of Torsades de Pointes" per www.crediblemeds.org/ that cannot be discontinued or replaced 7 days prior to starting study drug by safe alternative medication.•Inability to determine the QTcF interval
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g. uncontrolled diabetes, active or uncontrolled infection; uncontrolled arterial or pulmonary hypertension, uncontrolled clinically significant hyperlipidemia). Please refer to Section 6.3.1
* History of significant congenital or acquired bleeding disorder unrelated to cancer.
* Major surgery within 4 weeks prior to study entry or who have not recovered from prior surgery.
* History of other active malignancy within 3 years prior to study entry with the exception of previous or concomitant basal cell skin cancer and previous carcinoma in situ treated curatively
* History of acute pancreatitis within 1 year prior to randomization or medical history of chronic pancreatitis.
* History of chronic liver disease leading to severe hepatic impairment, or ongoing acute liver disease.
* Known hypersensitivity to the study treatment

Other protocol-defined Inclusion/exclusion criteria will apply.

Inclusion Criteria for optional TFR period:

Participants meeting the following additional criteria are not eligible to enter the TRI Period:

* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures
* A minimum of 5 years of study treatment up to maximum of 6 years of study treatment (i.e. participants are eligible to enter TFR any time between year 5 and year 6 of their study treatment
* Sustained MR 4.0 (BCR::ABL1 IS ≤0.01%) or better, assessed by central laboratory for at least 2 years (equivalent to 104 weeks) which includes MR 4.5 (BCR::ABL1 IS ≤0.0032%) for at least 1 year (equivalent to 52 weeks) immediately prior to entry into the TFR Period, with the 5 last consecutive RQ-PCR (every 12 weeks) assessments at/or below MR 4.5. Entry into TFR Period should be no later than 12 weeks from the last MR 4.5 RQ-PCR assessment
* Separate signed informed consent must be obtained prior to participation in the TFR Period

Exclusion Criteria for optional TFR period:

* Participants meeting the following additional criterion are not eligible for the inclusion in the optional TFR Period:
* Participants in the treatment re-initiation (TRI) Period cannot re-enter TFR for a second TFR attempt

Exclusion Criteria for Treatment Re-initiation (TRI) Period

Participants meeting the following additional criterion are not eligible to enter the TRI Period:

* In case of a pregnancy during the TFR Period, the pregnant woman must be discontinued upon loss of MMR (>0.1% BCR::ABL1 IS at a single assessment) and cannot enter the TRI Period
* Impaired cardiac function or cardiac repolarization abnormality
* Severe and/or uncontrolled concurrent medical disease that in the opinion of the Investigator could cause unacceptable safety risks or compromise compliance with the protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2028-01-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (106):
- United States (12):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists Pan, Tallahassee, Florida
  - University of Kentucky, Lexington, Kentucky
  - Uni of Massachusetts Medical Center, Worcester, Massachusetts
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Williamette Cancer Center, Eugene, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Avera Cancer, Sioux Falls, South Dakota
  - Chattanooga Onc And Hem Assoc PC, Chattanooga, Tennessee
  - Texas Oncology-Baylor USO, Dallas, Texas
  - Texas Oncology, Dallas, Texas
- Australia (4):
  - Novartis Investigative Site, Kingswood, New South Wales
  - Novartis Investigative Site, Port Macquarie, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Southport
- Novartis Investigative Site, Linz, Upper Austria, Austria
- Belgium (2):
  - Novartis Investigative Site, Leuven, Vlaams Brabant
  - Novartis Investigative Site, Brussels
- Novartis Investigative Site, Varna, Bulgaria
- Canada (4):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
- China (14):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Xian, Shanxi
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Lanzhou
  - Novartis Investigative Site, Tianjin
- Czechia (3):
  - Novartis Investigative Site, Ostrava, Poruba
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
- Denmark (2):
  - Novartis Investigative Site, Aarhus N
  - Novartis Investigative Site, Copenhagen
- Novartis Investigative Site, Helsinki, Finland
- France (4):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Germany (6):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Lübeck
- Hungary (3):
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Kaposvár
  - Novartis Investigative Site, Kecskemét
- Novartis Investigative Site, Delhi, India
- Israel (3):
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Verona, VR
- Japan (14):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Toyoake, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Chūō, Yamanashi
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Yamagata
- Malaysia (4):
  - Novartis Investigative Site, Kuantan, Pahang
  - Novartis Investigative Site, George Town, Pulau Pinang
  - Novartis Investigative Site, Subang Jaya, Selangor
  - Novartis Investigative Site, Kuala Selangor
- Novartis Investigative Site, Amsterdam, North Holland, Netherlands
- Norway (2):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Oslo
- Portugal (2):
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Vila Nova de Gaia
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Košice, Slovakia
- South Korea (2):
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Spain (5):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, El Palmar, Murcia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
- Novartis Investigative Site, Bellinzona, Switzerland
- Novartis Investigative Site, Taichung, Taiwan
- United Kingdom (3):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided are anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Hochhaus A, Wang J, Kim DW, Kim DDH, Mayer J, Goh YT, le Coutre P, Takahashi N, Kim I, Etienne G, Andorsky D, Issa GC, Larson RA, Bombaci F, Kapoor S, McCulloch T, Malek K, Yau L, Ifrah S, Hoch M, Cortes JE, Hughes TP; ASC4FIRST Investigators. Asciminib in Newly Diagnosed Chronic Myeloid Leukemia. N Engl J Med. 2024 Sep 12;391(10):885-898. doi: 10.1056/NEJMoa2400858. Epub 2024 May 31. PMID 38820078
- [Derived] Cortes JE, Hochhaus A, Takahashi N, Larson RA, Issa GC, Bombaci F, Ramscar N, Ifrah S, Hughes TP. Asciminib monotherapy for newly diagnosed chronic myeloid leukemia in chronic phase: the ASC4FIRST phase III trial. Future Oncol. 2022 Dec;18(38):4161-4170. doi: 10.2217/fon-2022-0923. Epub 2022 Dec 16. PMID 36524980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All trial participants randomized in a 1:1 ratio between asciminib and investigator selected TKI (imatinib 400 mg QD, nilotinib 300 mg BD, dasatinib 100 mg QD or bosutinib 400 mg QD).
Pre-assignment Details: Prior to randomization, the Investigator, in consultation with the participant, considering current treatment paradigm and participant characteristics - and comorbidities, made a selection of imatinib or 2G TKI (nilotinib, dasatinib, or bosutinib) to be used if the participant is randomized to the comparator arm.
  The enrolment into the strata of imatinib versus 2G TKI was managed by IRT to be approximately 50% versus 50%.
Groups:
- Asciminib (Imatinib Stratum): Patients took asciminib 80 mg QD under fasting conditions on ongoing basis.
- Asciminib (2nd Generation TKI Stratum): Patients took ascimimib 80 mg QD under fasting conditions on ongoing basis.
- Investigator Selected TKI (Imatinib Stratum): Patients took on ongoing basis the Investigator selected TKI (imatinib)
- Investigator Selected TKI (2nd Generation TKI Stratum: Patients took on ongoing basis the 2G investigator selected TKIs (nilotinib, or dasatinib, or bosutinib)
Period: Overall Study
Arm/Group | Asciminib (Imatinib Stratum) | Asciminib (2nd Generation TKI Stratum) | Investigator Selected TKI (Imatinib Stratum) | Investigator Selected TKI (2nd Generation TKI Stratum
Started | 101 | 100 | 102 | 102
Participants Not Treated | 1 | 0 | 2 | 1
Treated | 100 | 100 | 100 | 101
Completed (Participants for whom treatment is ongoing at the time of Data Cut-Off (DOC)) | 85 | 88 | 63 | 77
Not Completed | 16 | 12 | 39 | 25
Not completed — Unsatisfactory therapeutic effect | 6 | 6 | 21 | 10
Not completed — Adverse Event | 6 | 5 | 11 | 10
Not completed — Progressive disease | 2 | 0 | 3 | 1
Not completed — Protocol Deviation | 1 | 0 | 1 | 1
Not completed — Subject Decision | 0 | 1 | 1 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Participants not treated | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Investigator Selected TKI (2nd Generation TKI Stratum): Patients took on ongoing basis the 2G investigator selected TKIs (nilotinib, or dasatinib, or bosutinib)
- Total: Total of all reporting groups
Arm/Group | Asciminib (Imatinib Stratum) | Asciminib (2nd Generation TKI Stratum) | Investigator Selected TKI (Imatinib Stratum) | Investigator Selected TKI (2nd Generation TKI Stratum) | Total
Number analyzed (Participants) | 101 | 100 | 102 | 102 | 405
Age, Customized [Count of Participants; unit: Participants]
  18 to <65 years | 69 | 86 | 70 | 85 | 310
  65 to <75 years | 24 | 12 | 22 | 12 | 70
  >= 75 years | 8 | 2 | 10 | 5 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 31 | 37 | 42 | 149
  Male | 62 | 69 | 65 | 60 | 256
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 63 | 45 | 66 | 44 | 218
  Black or African American | 1 | 1 | 1 | 1 | 4
  Asian | 37 | 53 | 34 | 56 | 180
  Unknown | 0 | 1 | 1 | 1 | 3
EUTOS Long-Term Survival (ELTS) score [Count of Participants; unit: Participants] — ELTS score is a predictive and prognostic score used to estimate the risk of progression and survival risk in newly diagnosed patients with CML-CP.
  Participants
    Low | 62 | 60 | 64 | 61 | 247
    Intermediate | 30 | 26 | 30 | 27 | 113
    High | 9 | 14 | 8 | 14 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Molecular Response (MMR) at Week 48 - Ascimimib vs. Investigator Selected TKI
Description: Molecular response is assessed using BCR-ABL1 transcript levels measured by realtime quantitative polymerase chain reaction. MMR is defined as a ratio BCR-ABL/ABL ≤0.1% on the international scale (ie, at least 3 log reduction from a standardized baseline value).
Time Frame: At 48 weeks
Population: The Full Analysis Set (FAS) comprised of all participants to whom study treatment has been assigned by randomization.
Measure: Count of Participants; unit: Participants
Groups:
- Asciminib (All Asciminib ): Patients took asciminib 80 mg QD under fasting conditions on ongoing basis.
- Investigator Selected TKI (All Comparators): Patients took on ongoing basis the Investigator selected TKIs (imatinib, nilotinib, dasatinib or bosutinib)
Arm/Group | Asciminib (All Asciminib ) | Investigator Selected TKI (All Comparators)
Number analyzed (Participants) | 201 | 204
Participants | 136 | 100
Statistical Analysis 1: Comparison: Asciminib (All Asciminib ) vs Investigator Selected TKI (All Comparators); Test type: Superiority; p < 0.001, Mantel Haenszel; Risk Difference (RD) = 18.88, 95% CI 2-sided [9.59 to 28.17] — The Estimate Value is a percentage; The Confidence Interval are percentages

2. Secondary Outcome: Major Molecular Response at Week 96
Description: Molecular response is assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction. MMR is defined as a ratio BCR-ABL/ABL ≤0.1% on the international scale (ie, at least 3 log reduction from a standardized baseline value).
Time Frame: at 96 weeks (96 weeks after last patient first dose)
Reporting Status: Not Posted, anticipated posting 2028-10

3. Secondary Outcome: Time to Discontinuation of Study Treatment Due to Adverse Events (TTDAE)
Description: TTDAE is defined as the time from the date of first dose of study treatment to the date of discontinuation of study treatment due to Adverse Event (AE). For patients ongoing without study treatment discontinuation, on or prior to the analysis cut-off date, the time will be censored at the at the analysis cut-off date.
Time Frame: 96 weeks after last patient first dose
Reporting Status: Not Posted, anticipated posting 2028-10

4. Secondary Outcome: Major Molecular Response at Scheduled Data Collection Time Points
Description: as for outcome 2
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

5. Secondary Outcome: Major Molecular Response by Scheduled Data Collection Time Points
Description: as for outcome 2
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

6. Secondary Outcome: MR4.0 at Scheduled Data Collection Time Points
Description: Molecular response is assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction. MR4.0 is defined as a ratio BCR-ABL/ABL ≤0.01% on the international scale (ie, at least 4 log reduction from a standardized baseline value).
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

7. Secondary Outcome: MR4.5 at All Scheduled Data Collection Time Points
Description: Molecular response is assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction. MR4.5 is defined as a ratio BCR-ABL/ABL ≤0.0032% on the international scale (ie, at least 4.5 log reduction from a standardized baseline value).
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

8. Secondary Outcome: MR4.0 by Scheduled Data Collection Time Points
Description: as for outcome 6
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

9. Secondary Outcome: MR4.5 by All Scheduled Data Collection Time Points
Description: as for outcome 7
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

10. Secondary Outcome: Complete Hematological Response (CHR) at All Scheduled Data Collection Time Points
Description: Hematologic response will be assessed by CBC and physical examination at each visit.
  Complete Hematological Response (CHR) will be defined as all of the following present for ≥ 4 weeks:
  white blood cell(s) (WBC) count < 10 x 10^9/L PLT count < 450 x 10^9/L Basophils < 5% No blasts and promyelocytes in peripheral blood Myelocytes + metamyelocytes < 5% in peripheral blood No evidence of extramedullary disease, including spleen and liver
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

11. Secondary Outcome: Complete Hematological Response (CHR) by All Scheduled Data Collection Time Points
Description: as for outcome 10
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

12. Secondary Outcome: Percentage of Participants With Complete Cytogenic Response (CCyR) by Week 48 & Week 96
Description: The CCyR response status was to be based on bone marrow assessment. Bone marrow examination for cytogenetic assessment was to be performed locally by the Investigator at baseline for all participants. Thereafter, during the course of the study, cytogenetic assessment was not mandatory and only performed if clinically indicated.
Time Frame: By week 48 and by week 96 (48 weeks and 96 weeks after last patient first dose); data collection/analysis is ongoing for the 96 week time point, and the data will be reported later
Population: The Full Analysis Set (FAS) comprised of all participants to whom study treatment has been assigned by randomization and who had a valid bone marrow examination at week 48.
Measure: Count of Participants; unit: Participants
Groups:
- Investigator Selected TKI (All Comparators): Patients will take on ongoing basis the Investigator selected TKIs (imatinib, nilotinib, dasatinib or bosutinib)
Arm/Group | Asciminib (All Asciminib ) | Investigator Selected TKI (All Comparators)
Number analyzed (Participants) | 2 | 0
Participants
  Complete cytogenetic response (CCyR) | 1 | 0
  Partial cytogenetic response (PCyR) | 1 | 0
  Minor cytogenetic response (mCyR) | 0 | 0
  Minimal cytogenetic response | 0 | 0
  No cytogenetic response | 0 | 0

13. Secondary Outcome: Duration of MMR
Description: Duration of MMR is defined as the time between the date of the first documented achievement of MMR and the earliest date of loss of MMR, treatment failure, progression to Accelerated Phase/Blast Crisis, or CML-related death
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

14. Secondary Outcome: Duration of MR4.0
Description: Duration of MR4.0 is defined as the time between the date of the first documented achievement of MR4.0 and the earliest date of loss of MR4.0, treatment failure, progression to Accelerated Phase/Blast Crisis, or CML-related death
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

15. Secondary Outcome: Duration of MR4.5
Description: Duration of MR4.5 is defined as the time between the date of the first documented achievement of MR4.5 and the earliest date of loss of MR4.5, treatment failure, progression to Accelerated Phase/Blast Crisis, or CML-related death
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

16. Secondary Outcome: Time to First MMR
Description: Time to first MMR is defined as the time from the date of randomization to the date of the first documented occurrence of MMR. Time will be censored at the last molecular assessment date while on treatment, or the End Of Treatment (whichever comes first) for patients who have not experienced MMR.
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

17. Secondary Outcome: Time to First MR4.0
Description: Time to first MR4.0 is defined as the time from the date of randomization to the date of the first documented occurrence of MR4.0. Time will be censored at the last molecular assessment date while on treatment, or the End Of Treatment (whichever comes first) for patients who have not experienced MR4.0.
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

18. Secondary Outcome: Time to First MR4.5
Description: Time to first MR4.5 is defined as the time from the date of randomization to the date of the first documented occurrence of MR4.5. Time will be censored at the last molecular assessment date while on treatment, or the End Of Treatment (whichever comes first) for patients who have not experienced MR4.5.
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

19. Secondary Outcome: BCR-ABL1≤1% at Scheduled Data Collection Time Points
Description: Molecular response is assessed using BCR-ABL transcript levels measured by realtime quantitative polymerase chain reaction.
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

20. Secondary Outcome: BCR-ABL1≤1% by Scheduled Data Collection Time Points
Description: as for outcome 19
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

21. Secondary Outcome: Time to Treatment Failure (TTF)
Description: TTF is defined as the time from date of randomization to the first/earliest documented date of any of the following events: treatment failure as per ELN, Confirmed loss of MMR while on study treatment, discontinuation from study treatment due to any reason
  For patients that have not experienced an event prior to or at the analysis cut-off date, the time will be censored at the last study assessment date while on treatment, or the EOT (whichever comes first) .
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

22. Secondary Outcome: Failure Free Survival (FFS)
Description: FFS is defined as the time from the date of randomization to the earliest occurrence of the following events: treatment failure per ELN, confirmed loss of MMR, progression to AP/BC, death from any cause.
  For patients that have not experienced an event prior to or at the analysis cut-off date, the time will be censored at the date of last study treatment assessment or last post-treatment follow-up.
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

23. Secondary Outcome: Event Free Survival (EFS)
Description: EFS is defined as the time from the date of randomization to the earliest occurrence of the following events: treatment failure as per ELN, confirmed loss of MMR ,discontinuation of study treatment due to AE, progression to AP/BC, death from any cause.
  For patients that have not experienced an event prior to or at the analysis cut-off date, the time will be censored at the date of last study treatment assessment or last post-treatment follow-up.
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

24. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the earliest occurrence of progression to AP/BC or death from any cause.
  For patients that have not experienced an event prior to or at the analysis cut-off date, the time will be censored at the date of last study treatment assessment or last post-treatment follow-up.
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

25. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization to the date of death from any cause. For patients that have not experienced an event prior to or at the analysis cut-off date, the time will be censored at the date of last contact before the cut-off date.
Time Frame: Planned total follow-up duration of 5 years
Reporting Status: Not Posted, anticipated posting 2028-10

26. Secondary Outcome: Trough Plasma Concentrations.
Description: Trough plasma concentration will measure the concentration of asciminib in the blood immediately before the next dose is administered.
Time Frame: Week 48
Population: Pharmacokinetic analysis set (PAS): All participants to whom study treatment has been assigned by randomization to asciminib and that had a valid trough plasma concentration taken at week 48.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Asciminib (All Asciminib )
Number analyzed (Participants) | 107
ng/mL | 161 [11.9 to 1010]

27. Secondary Outcome: Pharmacokinetics (PK) of Asciminib: Cmax
Description: Cmax is the maximum serum concentration of asciminib during a dosing interval (mass x volume-1).
Time Frame: Week 2 (0 hours (h) pre-dose, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose)
Population: Full PK samples were collected at Week 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Asciminib (All Asciminib): Patients took asciminib 80 mg QD under fasting conditions on ongoing basis.
Arm/Group | Asciminib (All Asciminib)
Number analyzed (Participants) | 26
ng/mL | 1470 (38.2)

28. Secondary Outcome: PK of Asciminib: Tmax
Description: Tmax is the time to reach maximum (peak) plasma drug concentration after dose administration (time)
Time Frame: Week 2 (0 hours (h) pre-dose, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose)
Population: Full PK samples were collected at Week 2
Measure: Median (Full Range); unit: Hour (hr)
Arm/Group | Asciminib (All Asciminib)
Number analyzed (Participants) | 26
Hour (hr) | 2.00 [0.883 to 3.18]

29. Secondary Outcome: PK of Asciminib: AUCtau and AUClast
Description: AUCtau is the area under the plasma concentration-time curve over the dosing interval. AUClast is the area under the plasma concentration-time curve from time zero (time of dose administration) to time of last measurable concentration (mass x time x volume-1)
Time Frame: Week 2 (0 hours (h) pre-dose, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose)
Population: Full PK samples were collected at Week 2. Although samples were collected for 26 participants, AUCtau could not be evaluated because extrapolated AUC was over 20% for all participants.
  AUCtau is derived from extrapolated AUC. However, when it is over 20% for all participants, AUCtau cannot be determined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Asciminib (All Asciminib)
Number analyzed (Participants) | 26
ng*hr/mL
  AUClast | 8590 (42.2)
  AUCtau | NA (NA) — Although samples were collected for 26 participants, AUCtau could not be evaluated because extrapolated AUC was over 20% for all participants. AUCtau is derived from extrapolated AUC. However, when it is over 20% for all participants, AUCtau cannot be determined.

30. Secondary Outcome: PK of Asciminib: CL/F
Description: CL/F is the apparent total body clearance of asciminib from plasma after oral administration (volume x time-1).
Time Frame: Week 2 (0 hours (h) pre-dose, 1h, 2h, 3h, 4h, 6h, 8h and 12h post dose)
Population: Although samples were collected for 26 participants, CL/F could not be evaluated because extrapolated AUC was over 20% for all participants. CL/F is derived from extrapolated AUC. However, when it is over 20% for all participants, CL/F cannot be determined.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Asciminib (All Asciminib)
Number analyzed (Participants) | 26
ng*hr/mL | NA (NA) — Although samples were collected for 26 participants, CL/F could not be evaluated because extrapolated AUC was over 20% for all participants. CL/F is derived from extrapolated AUC. However, when it is over 20% for all participants, CL/F cannot be determined.

31. Secondary Outcome: Change From Baseline in Overall Scores (Global Health Status) and Individual Scales of the EORTC QLQ-C30 at Week 48 and Week 96
Description: The European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) assesses the quality of life of cancer patients. It consists of functioning scales, symptom scales, and the global health status quality of life (QoL) scale.
  A high score for functional and QoL items/scales from the QLQ-30 represents better function and QOL. A high score in symptoms items from QLQ-30 represents worse symptoms.
Time Frame: Baseline, week 48 and week 96
Population: Full Analysis Set: All participants who had an EORTC QLQ-C30 assessment both at baseline and at week 48.
Measure: Count of Participants; unit: Participants
Arm/Group | Asciminib (All Asciminib ) | Investigator Selected TKI (All Comparators)
Number analyzed (Participants) | 79 | 70
Participants
  Global health status/QoL: Very much better | 10 | 6
  Global health status/QoL: Moderately better | 18 | 7
  Global health status/QoL: A little better | 6 | 6
  Global health status/QoL: Unchanged | 28 | 26
  Global health status/QoL: A little worse | 5 | 6
  Global health status/QoL: Moderately worse | 10 | 12
  Global health status/QoL: Very much worse | 2 | 7
  Physical functioning: Very much better | 3 | 3
  Physical functioning: Moderately better | 10 | 12
  Physical functioning: A little better | 16 | 12
  Physical functioning: Unchanged | 32 | 26
  Physical functioning: A little worse | 7 | 8
  Physical functioning: Moderately worse | 10 | 6
  Physical functioning: Very much worse | 1 | 3
  Role functioning: Very much better | 5 | 7
  Role functioning: Moderately better | 10 | 7
  Role functioning: A little better | 0 | 0
  Role functioning: Unchanged | 54 | 41
  Role functioning: A little worse | 0 | 0
  Role functioning: Moderately worse | 4 | 7
  Role functioning: Very much worse | 6 | 8
  Emotional functioning: Very much better | 9 | 10
  Emotional functioning: Moderately better | 7 | 6
  Emotional functioning: A little better | 14 | 9
  Emotional functioning: Unchanged | 31 | 24
  Emotional functioning: A little worse | 7 | 10
  Emotional functioning: Moderately worse | 5 | 5
  Emotional functioning: Very much worse | 6 | 6
  Cognitive functioning: Very much better | 3 | 1
  Cognitive functioning: Moderately better | 13 | 8
  Cognitive functioning: A little better | 0 | 0
  Cognitive functioning: Unchanged | 44 | 36
  Cognitive functioning: A little worse | 0 | 0
  Cognitive functioning: Moderately worse | 16 | 19
  Cognitive functioning: Very much worse | 3 | 6
  Social functioning: Very much better | 7 | 6
  Social functioning: Moderately better | 14 | 6
  Social functioning: A little better | 0 | 0
  Social functioning: Unchanged | 51 | 40
  Social functioning: A little worse | 0 | 0
  Social functioning: Moderately worse | 4 | 7
  Social functioning: Very much worse | 3 | 11
  Fatigue: Very much better | 19 | 11
  Fatigue: Moderately better | 16 | 16
  Fatigue: A little better | 0 | 0
  Fatigue: Unchanged | 26 | 16
  Fatigue: A little worse | 0 | 0
  Fatigue: Moderately worse | 11 | 11
  Fatigue: Very much worse | 7 | 16
  Nausea and vomiting: Very much better | 1 | 1
  Nausea and vomiting: Moderately better | 7 | 5
  Nausea and vomiting: A little better | 0 | 0
  Nausea and vomiting: Unchanged | 67 | 48
  Nausea and vomiting: A little worse | 0 | 0
  Nausea and vomiting: Moderately worse | 3 | 11
  Nausea and vomiting: Very much worse | 1 | 5
  Pain: Very much better | 9 | 3
  Pain: Moderately better | 17 | 11
  Pain: A little better | 0 | 0
  Pain: Unchanged | 45 | 37
  Pain: A little worse | 0 | 0
  Pain: Moderately worse | 5 | 10
  Pain: Very much worse | 3 | 9
  Dyspnoea: Very much better | 11 | 9
  Dyspnoea: Moderately better | 0 | 0
  Dyspnoea: A little better | 0 | 0
  Dyspnoea: Unchanged | 59 | 49
  Dyspnoea: A little worse | 0 | 0
  Dyspnoea: Moderately worse | 0 | 0
  Dyspnoea: Very much worse | 9 | 12
  Insomnia: Very much better | 14 | 10
  Insomnia: Moderately better | 0 | 0
  Insomnia: A little better | 0 | 0
  Insomnia: Unchanged | 50 | 43
  Insomnia: A little worse | 0 | 0
  Insomnia: Moderately worse | 0 | 0
  Insomnia: Very much worse | 15 | 17
  Appetite loss: Very much better | 16 | 11
  Appetite loss: Moderately better | 0 | 0
  Appetite loss: A little better | 0 | 0
  Appetite loss: Unchanged | 59 | 51
  Appetite loss: A little worse | 0 | 0
  Appetite loss: Moderately worse | 0 | 0
  Appetite loss: Very much worse | 4 | 8
  Constipation: Very much better | 8 | 14
  Constipation: Moderately better | 0 | 0
  Constipation: A little better | 0 | 0
  Constipation: Unchanged | 58 | 40
  Constipation: A little worse | 0 | 0
  Constipation: Moderately worse | 0 | 0
  Constipation: Very much worse | 13 | 16
  Diarrhoea: Very much better | 11 | 8
  Diarrhoea: Moderately better | 0 | 0
  Diarrhoea: A little better | 0 | 0
  Diarrhoea: Unchanged | 61 | 43
  Diarrhoea: A little worse | 0 | 0
  Diarrhoea: Moderately worse | 0 | 0
  Diarrhoea: Very much worse | 7 | 19
  Financial difficulties: Very much better | 12 | 14
  Financial difficulties: Moderately better | 0 | 0
  Financial difficulties: A little better | 0 | 0
  Financial difficulties: Unchanged | 63 | 49
  Financial difficulties: A little worse | 0 | 0
  Financial difficulties: Moderately worse | 0 | 0
  Financial difficulties: Very much worse | 4 | 7

32. Secondary Outcome: Change From Baseline in EORTC QLQ-CML24 Scales at Week 48 and Week 96
Description: The QLQ-CML24 consists of multi-scale items: symptom burden, impact on worry/mood, impact on daily life, body image problems, satisfaction with care and information and satisfaction with social life.
  A higher score on most of the item scales in QLQ-CML24 reflects a larger impairment in the corresponding domain, with the exception of the satisfaction with care and information, and problems and satisfaction with social life, where a higher score reflects a higher level of satisfaction.
Time Frame: Baseline, week 48 and week 96.
Population: Full Analysis Set: All participants who had an EORTC QLQ-CML24 assessment both at baseline and at week 48.
Measure: Count of Participants; unit: Participants
Arm/Group | Asciminib (All Asciminib) | Investigator Selected TKI (All Comparators)
Number analyzed (Participants) | 77 | 66
Participants
  Symptom Burden: Very much better | 0 | 2
  Symptom Burden: Moderately better | 12 | 4
  Symptom Burden: A little better | 18 | 5
  Symptom Burden: Unchanged | 27 | 22
  Symptom Burden: A little worse | 7 | 16
  Symptom Burden: Moderately worse | 6 | 12
  Symptom Burden: Very much worse | 7 | 5
  Impact on Worry/Mood: Very much better | 11 | 7
  Impact on Worry/Mood: Moderately better | 7 | 9
  Impact on Worry/Mood: A little better | 20 | 6
  Impact on Worry/Mood: Unchanged | 17 | 18
  Impact on Worry/Mood: A little worse | 16 | 11
  Impact on Worry/Mood: Moderately worse | 2 | 4
  Impact on Worry/Mood: Very much worse | 4 | 11
  Impact on Daily Life: Very much better | 21 | 17
  Impact on Daily Life: Moderately better | 26 | 10
  Impact on Daily Life: A little better | 0 | 0
  Impact on Daily Life: Unchanged | 19 | 23
  Impact on Daily Life: A little worse | 0 | 0
  Impact on Daily Life: Moderately worse | 6 | 5
  Impact on Daily Life: Very much worse | 5 | 11
  Body Image Problems: Very much better | 18 | 10
  Body Image Problems: Moderately better | 0 | 0
  Body Image Problems: A little better | 0 | 0
  Body Image Problems: Unchanged | 48 | 41
  Body Image Problems: A little worse | 0 | 0
  Body Image Problems: Moderately worse | 0 | 0
  Body Image Problems: Very much worse | 11 | 15
  Satisfaction with Care and Information: Very much better | 8 | 13
  Satisfaction with Care and Information: Moderately better | 5 | 4
  Satisfaction with Care and Information: A little better | 0 | 0
  Satisfaction with Care and Information: Unchanged | 30 | 31
  Satisfaction with Care and Information: A little worse | 0 | 0
  Satisfaction with Care and Information: Moderately worse | 18 | 7
  Satisfaction with Care and Information: Very much worse | 16 | 11
  Satisfaction with Social Life: Very much better | 15 | 14
  Satisfaction with Social Life: Moderately better | 0 | 0
  Satisfaction with Social Life: A little better | 0 | 0
  Satisfaction with Social Life: Unchanged | 40 | 37
  Satisfaction with Social Life: A little worse | 0 | 0
  Satisfaction with Social Life: Moderately worse | 0 | 0
  Satisfaction with Social Life: Very much worse | 22 | 15

33. Primary Outcome: Percentage of Participants With Major Molecular Response (MMR) at Week 48 - Asciminib (Imatinib Stratum) vs Investigator Selected TKI (Imatinib Stratum)
Description: Molecular response is assessed using BCR-ABL1 transcript levels measured by realtime quantitative polymerase chain reaction. MMR is defined as a ratio BCR-ABL1/ABL ≤0.1% on the international scale (ie, at least 3 log reduction from a standardized baseline value).
Time Frame: At 48 weeks
Population: The IMA Full Analysis Set (FASIMA) comprised of all participants from the FAS, whose PRS TKI is imatinib. FAS comprised of all participants to whom study treatment has been assigned by randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Asciminib (Imatinib Stratum) | Investigator Selected TKI (Imatinib Stratum)
Number analyzed (Participants) | 101 | 102
Participants | 70 | 41
Statistical Analysis 1: Comparison: Asciminib (Imatinib Stratum) vs Investigator Selected TKI (Imatinib Stratum); Test type: Superiority; p < 0.001, Mantel Haenszel; Risk Difference (RD) = 29.55, 95% CI 2-sided [16.91 to 42.18] — The Estimate Value is a percentage; The Confidence Interval are percentages

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are collected from first dose of study treatment until end of study treatment plus 30 days post treatment. AEs reported in this record are from first dose of study treatment until data cut-off on 28-Nov-2023 (approx. 2 years).
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- Imatinib: Patients took on ongoing basis the Investigator selected TKI (imatinib).
- 2nd Generation TKI: Patients took on ongoing basis the 2nd Generation investigator selected TKIs (nilotinib, or dasatinib, or bosutinib)
- All Comparators: Patients took on ongoing basis the Investigator selected TKIs (imatinib, nilotinib, dasatinib or bosutinib)
Arm/Group | Asciminib (All Asciminib) | Imatinib | 2nd Generation TKI | All Comparators
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/99 | 0/102 | 0/201
Serious Adverse Events (participants affected / at risk) | 22/200 | 12/99 | 20/102 | 32/201
Other Adverse Events (participants affected / at risk) | 177/200 | 89/99 | 100/102 | 189/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asciminib (All Asciminib) (N=200) | Imatinib (N=99) | 2nd Generation TKI (N=102) | All Comparators (N=201)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0
Epiretinal membrane (Eye disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Budd-Chiari syndrome (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Alveolar osteitis (Infections and infestations) | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 2
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 2
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1
Device dislocation (Product Issues) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Asciminib (All Asciminib) (N=200) | Imatinib (N=99) | 2nd Generation TKI (N=102) | All Comparators (N=201)
Anaemia (Blood and lymphatic system disorders) | 23 | 26 | 23 | 49
Leukopenia (Blood and lymphatic system disorders) | 16 | 12 | 7 | 19
Neutropenia (Blood and lymphatic system disorders) | 21 | 15 | 16 | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 14 | 17 | 31
Vertigo (Ear and labyrinth disorders) | 1 | 5 | 4 | 9
Dry eye (Eye disorders) | 11 | 4 | 4 | 8
Eyelid oedema (Eye disorders) | 0 | 8 | 0 | 8
Periorbital oedema (Eye disorders) | 2 | 10 | 1 | 11
Abdominal pain (Gastrointestinal disorders) | 16 | 3 | 9 | 12
Constipation (Gastrointestinal disorders) | 19 | 4 | 12 | 16
Diarrhoea (Gastrointestinal disorders) | 31 | 26 | 26 | 52
Dyspepsia (Gastrointestinal disorders) | 5 | 5 | 5 | 10
Nausea (Gastrointestinal disorders) | 18 | 21 | 18 | 39
Vomiting (Gastrointestinal disorders) | 11 | 12 | 6 | 18
Asthenia (General disorders) | 8 | 8 | 3 | 11
Face oedema (General disorders) | 0 | 10 | 0 | 10
Fatigue (General disorders) | 28 | 14 | 18 | 32
Oedema peripheral (General disorders) | 3 | 7 | 6 | 13
Pyrexia (General disorders) | 10 | 6 | 3 | 9
COVID-19 (Infections and infestations) | 35 | 18 | 20 | 38
Herpes zoster (Infections and infestations) | 3 | 6 | 0 | 6
Nasopharyngitis (Infections and infestations) | 12 | 6 | 5 | 11
Upper respiratory tract infection (Infections and infestations) | 14 | 9 | 7 | 16
Alanine aminotransferase increased (Investigations) | 14 | 6 | 19 | 25
Amylase increased (Investigations) | 10 | 4 | 6 | 10
Aspartate aminotransferase increased (Investigations) | 4 | 6 | 15 | 21
Blood alkaline phosphatase increased (Investigations) | 11 | 13 | 6 | 19
Blood bilirubin increased (Investigations) | 5 | 2 | 11 | 13
Blood creatine phosphokinase increased (Investigations) | 9 | 4 | 6 | 10
Blood creatinine increased (Investigations) | 3 | 5 | 4 | 9
Gamma-glutamyltransferase increased (Investigations) | 13 | 4 | 9 | 13
Lipase increased (Investigations) | 22 | 14 | 11 | 25
Lymphocyte count decreased (Investigations) | 10 | 12 | 3 | 15
Neutrophil count decreased (Investigations) | 29 | 16 | 21 | 37
Platelet count decreased (Investigations) | 29 | 14 | 18 | 32
White blood cell count decreased (Investigations) | 22 | 17 | 13 | 30
Decreased appetite (Metabolism and nutrition disorders) | 5 | 4 | 6 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 7 | 3 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 6 | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 8 | 7 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 9 | 9 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 19 | 5 | 24
Myalgia (Musculoskeletal and connective tissue disorders) | 26 | 17 | 15 | 32
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 6 | 4 | 10
Dizziness (Nervous system disorders) | 8 | 2 | 6 | 8
Headache (Nervous system disorders) | 26 | 8 | 22 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 6 | 10 | 16
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 4 | 9 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 0 | 7 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 4 | 3 | 7
Rash (Skin and subcutaneous tissue disorders) | 26 | 10 | 22 | 32
Hypertension (Vascular disorders) | 14 | 6 | 2 | 8

LIMITATIONS AND CAVEATS:
Adverse Events data were not collected from the 4 participants who are not included in the Safety Set as they did not receive any treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT04971226/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/26/NCT04971226/SAP_001.pdf